CLINICAL TRIAL: NCT01155232
Title: Effect of 24 Months of Teriparatide Therapy on Bone Microarchitecture and Bone Volume in Men and Women With Osteoporosis
Brief Title: Effects of Teriparatide (PTH) on Bone in Men and Women With Osteoporosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 04-0655
Record Dates: First submitted 2010-06-29; First posted 2010-07-01 (Estimated); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Osteoporosis
Keywords: osteoporosis; Forteo; Parathyroid hormone; HR-pQCT
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Forteo (teriparatide): postmenopausal women and men with osteoporosis Teriparatide is marketed as Forteo by Eli Lilly Teriparatide is not supplied (observational study)
  Interventions: Drug: Teriparatide
- Forteo (teriparatide) in AFF: women who have experienced an atypical femur fracture (AFF) Teriparatide is not supplied (observational study)
  Interventions: Drug: Teriparatide

INTERVENTIONS:
Drug: Teriparatide — Forteo (teriparatide)pen daily for 24 months
  Other Names: Teriparatide is a section of the parathyroid hormone (PTH) given by injection.; The drug is marketed by Eli Lilly under the name of Forteo

SUMMARY:
Teriparatide (PTH) is the only bone formation therapy that has been approved for the treatment of postmenopausal osteoporosis in Canada. Osteoporosis is currently diagnosed using a bone mineral density (BMD) scan, which measures the amount of mineral (calcium etc) in bones (the higher the amount of mineral, the lower the fracture risk). Although BMD is linked to bone strength and is used to measure fracture risk, it does not give information on bone structure (called bone geometry) which can also tell us a great deal about fracture risks. Clinical trials have shown that teriparatide increases BMD at the lumbar spine and total hip, while BMD at the forearm may decrease after 20 months of therapy. However, bone biopsies of the pelvis done on people taking teriparatide show improvement of bone geometry (ie bone thickness and increased trabeculae (small interconnecting rods of bone), suggesting that a change in bone geometry at the wrist may be occurring as well. Currently, there is a new technology, high resolution pQCT (HR-pQCT) that can assess bone geometry without a biopsy. Since bone strength is affected both by BMD and bone structure (as well as other material properties), our group is interested in examining changes in bone geometry at the radius and tibia in men and women with osteoporosis who receives 24 months of teriparatide therapy.

The investigators believe that this new approach of measuring bone strength will help us better understand the mechanisms of therapeutic efficacy of teriparatide. In addition, measuring indices of bone strength such as the material composition (bone mineral content or BMD) and structural properties of bone (size and shape, and microarchitecture) may provide more data about the mechanisms of how teriparatide treatment can decrease fracture risk. In the end, this data will benefit and improve patient care by allowing us to show patients and their providers that whether BMD increases, decreases or stay the same, there are changes in their bone geometric structure with teriparatide therapy that increases bone strength.

DETAILED DESCRIPTION:
Teriparatide (PTH) is the only bone formation therapy that has been approved for the treatment of postmenopausal osteoporosis in Canada. Randomized controlled trials have shown that teriparatide increases bone mineral density (BMD) at the lumbar spine and total hip, while BMD at the forearm may decrease after 20 months of therapy. It is believed that the decline in BMD at the distal radius observed during teriparatide therapy may not be indicative of decreases in bone strength, but may be a result of increases in the width of the radius. Teriparatide works by inducing new periosteal bone apposition, which results in improved bone geometry and increased bone strength that may not be reflected by BMD measurements. However, there is no published data on bone geometric changes at the radius either by bone biopsy or by HR-pQCT in patients receiving teriparatide therapy. It is our intention to fill this gap in knowledge with regard to how teriparatide affects BMD and bone structure at the radius and tibia in men and women with osteoporosis.

The main objectives of this study are to determine the effect of 24 months of teriparatide therapy on cortical thickness, trabecular thickness, trabecular number, trabecular separation and BV/TV, as measured by HR-pQCT (XtremeCT, Scanco Medical, Switzerland) at the radius and tibia in men and women with osteoporosis. The primary outcome will be cortical thickness; the other measures will be secondary outcomes. The secondary objective is to determine the effect of 24 months of teriparatide therapy on moment of inertia, connectivity index, and bone strength, as measured by the HR-pQCT and calculated using finite element modeling analysis at the radius and tibia in men and women with osteoporosis.

This is an open label before and after study of a cohort of 100 men and women taking teriparatide for 24 months. As this is an observational study, study medication will not be supplied to study participants.

Recruitment of these subjects will be by referral from specialty clinics of the participating investigators. Participants will undergo two (2) procedures on five (7) separate occasions (at baseline, 6, 12, 18 and at 24 months, and then post therapy at 36 and 48 months). The procedures are HR-pQCT and DXA. In addition to the above procedures, subjects will be asked to complete blood tests which are part of standard clinical practice. Blood will be done both at baseline, 1 month and at 18 month. A follow up phone call will also be made to the patient at 1 month to discuss any updates in patient's health status and to ensure that patients complete the 1 month blood tests.

Understanding the effect of teriparatide on bone geometry and BMD will enable us to better understand the effect of teriparatide on bone strength at the radius and the tibia, and bone strength in general, even when the BMD stays the same or decreases after a course of treatment.

ELIGIBILITY:
Inclusion Criteria:

* History of fragility fracture OR
* High risk for fractures OR
* Very low BMD (T-score ≤ -2.5) OR
* Failed or intolerant to bisphosphonates
* Baseline serum levels of calcium, urate, ALP, PTH, creatinine and 25- hydroxyvitamin D [25(OH)D] must be within acceptable normal limits
* Ability to obtain teriparatide (not supplied by study sponsor)

Exclusion Criteria:

* History of skeletal irradiation
* Those at increased risk for osteosarcoma
* Diagnosis of Paget's disease
* History of primary hyperparathyroidism
* Significant renal impairment
* Vitamin D deficiency
* On steroids or have other causes of secondary osteoporosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: community dwelling men and women with osteoporosis who have been prescribed teriparatide for severe osteoporosis. (Teriparatide is not supplied as part of this study)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2004-11; Primary Completion 2025-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in cortical thickness at the radius and tibia as measured by high-resolution quantitative computer tomography (HR-pQCT) | 0-24 months

CONTACTS AND LOCATIONS:
Overall Officials: Angela m Cheung, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, TGH, Toronto, Ontario, Canada